CLINICAL TRIAL: NCT00757926
Title: Phase I/II, Randomized, Double-blind, Placebo-controlled, Staged Dosage Escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity of a 3-dose Series of Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine [BRV-TV] Administered to Healthy Indian Infants Concurrently With Other Standard EPI Vaccines
Brief Title: Safety and Immunogenicity Study of the Recombinant Human Bovine Reassortant Rotavirus Vaccine in Healthy Indian Infants
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Replaced with an alternate study
Sponsor: Shantha Biotechnics Limited (Industry)
Collaborators: PATH (Other)
Responsible Party: Dr. Raman Rao, Head clinical Research and Medical Affairs, Shantha Biotechnics Limited, Hyderabad
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: SBL/BRV-TV/PhI/2008/0100
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Rotavirus Infections
MeSH Terms: conditions — Rotavirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Biological: Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine [BRV-TV]
- 2 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine [BRV-TV] — Three oral doses of the vaccine (0.5 ml each) following oral administration of antacid.
  Arms: 1
Other: Placebo — Three oral doses of the placebo (0.5 ml each)following oral administration of antacid.
  Arms: 2

SUMMARY:
A randomized, double-blind, placebo-controlled, staged dosage escalation study to evaluate the safety, tolerability, and immunogenicity of a 3-dose series of Live Attenuated Tetravalent (G1-G4) Bovine-Human Reassortant Rotavirus Vaccine [BRV-TV] administered to healthy Indian infants concurrently with other standard EPI vaccines would be undertaken to evaluate the study hypothesis that a 3-dose series of BRV-TV (containing the VP7 serotypes G1, G2, G3, and G4) administered orally to healthy Indian infants at 6-8, 10-12, and 14-16 weeks of age concurrently with other standard EPI vaccines would be generally well tolerated and immunogenic.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants 6-8 weeks of age of either sex;
* Born after a gestational period of 36-42 weeks with birth weight >2 kg;
* Father, mother or other legally acceptable representative (guardian) properly informed about the study and having signed the informed consent form (ICF);
* Parent or guardian available for the entire period of the study and reachable by study staff for post-vaccination follow-up.

Exclusion Criteria:

* History of congenital abdominal disorders, intussusception, or abdominal surgery;
* Known or suspected impairment of immunological function;
* Known hypersensitivity to any component of the rotavirus vaccine;
* Prior receipt of any rotavirus vaccine;
* Fever, with an oral temperature ≥38.1oC (≥100.5oF); presumably measured by study staff?
* History of known rotavirus disease, chronic diarrhea, or failure to thrive;
* Baseline level of ALT or AST >2.5 times the upper limit of normal;
* Clinical evidence of active gastrointestinal illness (infants with GERD can participate in the study so long as this condition is well controlled with or without medication);
* Receipt of any IM, oral, or IV corticosteroid treatment (infants on inhaled steroids may be permitted to participate in the study);
* Infants residing in a household with an immuno-compromised person (e.g., individuals with a congenital immunodeficiency, HIV infection, leukemia, lymphoma, Hodgkin's disease, multiple myeloma, generalized malignancy, chronic renal failure, nephrotic syndrome, organ or bone marrow transplantation, or those receiving immunosuppressive chemotherapy including long-term systemic corticosteroids);
* Infants testing positive for HBV, HCV, or HIV infection;
* Prior receipt of a blood transfusion or blood products, including immunoglobulins;
* Any infants who can not be adequately followed for safety by telephone and/or a home visit;
* Any conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 240 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-08 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Upto one month after each of the three doses of vaccine/ placebo

SECONDARY OUTCOMES:
Immunogenicity | At one month after each of the three doses of vaccine/ placebo
Viral Shedding | After each of the three doses of the vaccine/placebo

CONTACTS AND LOCATIONS:
Overall Officials: Raman Rao, MD, Study Director — Shantha Biotechnics Limited
Locations (1):
- Christian Medical College, Vellore, Tamil Nadu, India